CLINICAL TRIAL: NCT02451228
Title: Pharmacokinetic and Pharmacogenomic Approach to Indomethacin Therapy in Pregnancy
Brief Title: Indomethacin PK and PD Therapy in Pregnancy
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-0067; 1R01HD083003-01 (NIH)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2018-02

CONDITIONS: Premature Labor; Pregnancy; Premature Birth
Keywords: Pharmacokinetics; Pharmacodynamics; Preterm labor; Preterm birth; Estradiol; Indomethacin; Pregnancy; Short Cervix; CYP2C9 Genotype
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal Venous Blood for serum Maternal Blood for DNA (for CYP2C9) Maternal Urine Cord Blood (Umbilical Vein and Artery) for serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group: Observational opportunistic pharmacokinetic study of 300 pregnant women receiving Indomethacin therapy as standard of care for risk of preterm birth. Receive serial blood collection from IV.
  Interventions: Other: Serial blood collection

INTERVENTIONS:
Other: Serial blood collection — Serial blood collection from IV for pharmacokinetic and pharmacodynamic analysis. No drug, device, or biologic intervention. Opportunistic.

SUMMARY:
This study will follow pregnant women who are taking indomethacin as Standard of Care (SOC) for the indications of preterm labor (PTL), short cervix, or other indications, to evaluate the pharmacokinetics (PK), what the body does to the drug, and pharmacodynamics (PD), effectiveness of the drug in treating the specific intended disease process of this medication. This will help us develop more information for medication dosing specific to pregnant women experiencing preterm labor.

Indomethacin is often prescribed to pregnant women presenting with preterm labor or shortened cervix, which places them at risk for preterm labor and delivery. Indomethacin has been used since the 1970s to prolong pregnancy by decreasing uterine contractions. However, despite the widespread use of indomethacin in pregnancy, there is limited information available to help physicians determine how much indomethacin to prescribe and how often to prescribe it.

DETAILED DESCRIPTION:
Opportunistic study of indomethacin prescribed to patients per standard of care. Determine the pharmacokinetics, pharmacodynamics and pharmacogenomics of Indomethacin in pregnant patients with the hypothesis that that estradiol levels during pregnancy (12-32 weeks of gestation) and CYP2C9 polymorphisms affect the PK of indomethacin, and subsequently, the response to indomethacin therapy in patients at risk of Preterm birth (PTB). This hypothesis will be tested with the following specific aims: (1) Determine the PK of indomethacin in pregnant women at risk of PTB and its PD effects on reducing the rate of PTB before 34 weeks of gestation, as well as any associations between the PK and secondary maternal/neonatal clinical outcomes; (2) Determine the effects of maternal levels of estradiol in mid-pregnancy and CYP2C9 polymorphisms on indomethacin biotransformation to O-desmethylindomethacin in pregnant patients; (3) Construct a population PK/PD model of indomethacin in patients at risk of PTB (12-32 weeks of gestation) in order to optimize the dose and the dosing frequency for indomethacin prescribed to each individual based on covariates such as race/ethnicity, CYP2C9 genotype, gestational age, estradiol levels, smoking status, and body mass index (BMI). The investigators will enroll 300 subjects with spontaneous preterm labor (sPTL) or shortened cervix in a prospective opportunistic PK study designed to correlate the PK of indomethacin, patient genotype, and clinical outcomes. The investigators will merge dosing, sampling, demographic, and clinical information with the drug concentration data and use population PK methodologies to analyze the data using nonlinear mixed effect modeling. Quantification of the differences within and between individuals allows for identification of covariates (e.g., CYP2C9 genotype, estradiol levels, BMI, etc.) that can explain variability and affect drug exposure. These covariates, if significant, can then be used in the future to optimize dosing in individual patients at risk for PTB. Achieving this goal of individualized indomethacin therapy could have a significant impact on clinical practice and improve maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, patients must meet all of the following criteria:

1. Age at least 18 years
2. Singleton gestation
3. 12 0/7 to 32 0/7 weeks gestation (see Gestational Age Determination section 3.2.1.1)
4. Patient receiving indomethacin for any of the following diagnoses:

   1. Preterm labor: regular uterine contractions with documented cervical change or dilatation ≥ 2 cm and 80% effacement
   2. Cervical shortening (< 2.5 cm documented on transvaginal ultrasound) with or without funneling membranes
   3. Planned cervical cerclage or emergent cerclage
   4. Other condition whereby Indomethacin is indicated
5. Maternal and fetal condition allows anticipated delay of delivery for more than 24 hours -

Exclusion Criteria:

* Exclusion criteria include:

  1. Contraindications to indomethacin use (history of maternal bleeding disorder, thrombocytopenia, maternal hepatic, gastrointestinal ulcerative, or renal dysfunction, asthma)
  2. Known fetal abnormality, genetic syndrome, or intrauterine fetal demise
  3. Anticipated delivery in less than 24 hours, cervical dilatation > 6 cm
  4. Preterm premature rupture of membranes
  5. Suspected chorioamnionitis
  6. Oligohydramnios (DVP < 2 cm)
  7. Congenital Uterine anomaly
  8. Vaginal bleeding due to suspected placental abruption or placenta previa
  9. Planned preterm delivery for maternal/fetal indications
  10. Non-reassuring fetal status
  11. Planned delivery outside UTMB or participation in another intervention trial which may affect maternal or neonatal outcomes
  12. Unsure gestational age due to possibility of intrauterine growth restriction
  13. Hematocrit <28% (as determined by most recent result within 1 month of enrollment)
  14. Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi-center study including 300 pregnant women between 12-32 weeks of gestation at risk of PTB (sPTL or shortened cervix with or without funneling membranes) or other conditions to whom indomethacin is prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2015-05; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Gestational age at delivery | Enrollment until delivery of the participant
  Gestational age at delivery calculated from the first day of last menstrual period unless "unsure" and then it will be calculated from ultrasound measurements

SECONDARY OUTCOMES:
Maternal outcomes | Enrollment until delivery and maternal discharge
  Diagnosed maternal outcomes including oligohydramnios, chorioamnionitis, preterm premature rupture of membranes, venous thromboembolism, pulmonary edema, postpartum hemorrhage, and maternal death
Neonatal outcomes | The earlier of neonatal discharge or up to 120 days postnatal
  Diagnosed neonatal outcomes including birth weight, APGAR scores, neonatal sepsis, respiratory distress syndrome, patent ductus arteriosis, necrotizing enterocolitis, broncopulmonary dysplasia, paraventricular leukomalacia, intraventricular hemorrhage, fetal, or neonatal death
Neonatal admission to Neonatal intensive care unit (NICU) | The earlier of neonatal discharge or up to 120 days postnatal
  Documentation of NICU admission [yes/no]
Length of stay in the Neonatal intensive care unit (NICU) | The earlier of neonatal discharge or up to 120 days postnatal
  If admitted to the NICU, number of days in the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hankins, MD, Principal Investigator — University of Texas; Erik Rytting, PhD, Principal Investigator — University of Texas
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - University of Texas Medical Branch, Dept of OB/GYN, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Once published